CLINICAL TRIAL: NCT05504265
Title: Comparison of Efficacy and Safety of Different Analgesic Modes in Minimally Invasive Esophagectomy for Esophageal Cancer
Brief Title: Perioperative Analgesia Modes in Minimally Invasive Esophagectomy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22/166-3367
Record Dates: First submitted 2022-07-18; First posted 2022-08-17 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Cancer; Perioperative Analgesia; NSAIDs; Opioid; Patient-controlled Analgesia
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Postoperative NSAIDs (Other)
  Interventions: Drug: Postoperative flurbiprofen axetil
- Preemptive analgesia followed by Postoperative NSAIDs (Experimental)
  Interventions: Drug: Preemptive flurbiprofen axetil; Drug: Postoperative flurbiprofen axetil
- Postoperative patient-controlled analgesia pump (Experimental)
  Interventions: Device: Patient-controlled analgesia pump

INTERVENTIONS:
Drug: Preemptive flurbiprofen axetil — 50mg once，30min before induction anesthesia
  Arms: Preemptive analgesia followed by Postoperative NSAIDs
Drug: Postoperative flurbiprofen axetil — 50mg bid
  Arms: Postoperative NSAIDs; Preemptive analgesia followed by Postoperative NSAIDs
Device: Patient-controlled analgesia pump — Sufentanil 2.5 μg/kg+ondansetron 8mg, prepared to 100ml normal saline; background dose: 2 ml/h, single press analgesic pump injection volume: 0.5 ml, locking time: 15 min.
  Arms: Postoperative patient-controlled analgesia pump

SUMMARY:
This study was designed to compare analgesic efficacy and safety of different perioperative analgesic modes in minimally invasive esophagectomy for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years;
* Patients underwent laparoscopic and thoracoscopic or robotic-assisted minimally invasive esophagectomy ;
* Informed consent.

Exclusion Criteria:

* Has a history of cholecystitis or urolithiasis within 3 months;
* Has a history of atherothrombosis (peripheral arterial disease), stroke, myocardial infarction;
* With lung diseases, such as pneumonia, atelectasis, emphysema, pulmonary bullae, etc;
* Preoperative cardiac function grade ≥ III or coronary artery stenosis;
* Preoperative indwelling of a thoracic drainage tube;
* Long-term heavy drinker(heavy drinking was defined as follows: for men, consuming more than 4 drinks on any day or more than 14 drinks per week; For women, consuming more than 3 drinks on any day or more than 7 drinks per week);
* Opioid-tolerant patients(defined as those who have been taking, for a week or longer, at least 60 mg of morphine daily, or at least 30 mg of oral oxycodone daily, or at least 8 mg of oral hydromorphone daily or an equianalgesic dose of another opioid);
* With painful skin complications, such as rashes and blisters;
* Conversion to open surgery;
* The postoperative ventilation function was limited, or the duration of endotracheal intubation was more than 24h.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain score | 4 hours after surgery
  In the Visual Analog Score to be used as the pain measurement criterion, '0' is the minimum value that indicates no pain, while '10' is the maximum value that defines the most severe pain.
Postoperative pain score | 12 hours after surgery
  In the Visual Analog Score to be used as the pain measurement criterion, '0' is the minimum value that indicates no pain, while '10' is the maximum value that defines the most severe pain.
Postoperative pain score | 24 hours after surgery
  In the Visual Analog Score to be used as the pain measurement criterion, '0' is the minimum value that indicates no pain, while '10' is the maximum value that defines the most severe pain.
Postoperative pain score | 36 hours after surgery
  In the Visual Analog Score to be used as the pain measurement criterion, '0' is the minimum value that indicates no pain, while '10' is the maximum value that defines the most severe pain.
Postoperative pain score | 48 hours after surgery
  In the Visual Analog Score to be used as the pain measurement criterion, '0' is the minimum value that indicates no pain, while '10' is the maximum value that defines the most severe pain.
Postoperative pain score | 60 hours after surgery
  In the Visual Analog Score to be used as the pain measurement criterion, '0' is the minimum value that indicates no pain, while '10' is the maximum value that defines the most severe pain.
Postoperative pain score | 72 hours after surgery
  In the Visual Analog Score to be used as the pain measurement criterion, '0' is the minimum value that indicates no pain, while '10' is the maximum value that defines the most severe pain.

SECONDARY OUTCOMES:
Time to first postoperative flatus | Up to 14 days after surgery
  Time from the end of surgery to the first flatus.
Time to first postoperative defaecation | Up to 14 days after surgery
  Time from the end of surgery to the first defaecation.
Abdominal distension score | 24 hours after surgery
  Abdominal distension was measured using a scoring system, '0' is the minimum value that indicates no abdominal distension, while '10' is the maximum value that defines the most severe abdominal distension.
Abdominal distension score | 48 hours after surgery
  Abdominal distension was measured using a scoring system, '0' is the minimum value that indicates no abdominal distension, while '10' is the maximum value that defines the most severe abdominal distension.
Abdominal distension score | 72 hours after surgery
  Abdominal distension was measured using a scoring system, '0' is the minimum value that indicates no abdominal distension, while '10' is the maximum value that defines the most severe abdominal distension.
Side effects related to opioids | 24 hours after surgery
  Nausea and vomiting were measured using a scoring system(0 = no nausea, 1 = only nausea, 2 = both nausea and vomiting).
Side effects related to opioids | 48 hours after surgery
  Nausea and vomiting were measured using a scoring system(0 = no nausea, 1 = only nausea, 2 = both nausea and vomiting).
Side effects related to opioids | 72 hours after surgery
  Nausea and vomiting were measured using a scoring system(0 = no nausea, 1 = only nausea, 2 = both nausea and vomiting).
Time to first postoperative ambulation | Up to 14 days after surgery
  Time from the end of surgery to the first postoperative ambulation
Hospital duration from operation to discharge | Up to 60 days after surgery
  Time from the end of surgery to discharge from the hospital
Rate of pulmonary infection | Up to 30 days after surgery
  Rate of pulmonary infection up to 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No